CLINICAL TRIAL: NCT06803875
Title: A Phase 1/2 Study of hALK.CAR T Cells for Patients With Relapsed/Refractory High-risk Neuroblastoma
Brief Title: Study of hALK.CAR T Cells for Patients With Relapsed/Refractory High-risk Neuroblastoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Roberto Chiarle (Other)
Collaborators: Boston Children's Hospital (Other); Dana-Farber Cancer Institute (Other)
Responsible Party: Sponsor-Investigator, Roberto Chiarle, Professor in Pathology, Boston Children's Hospital
Organization: Boston Children's Hospital (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 24-392
Record Dates: First submitted 2024-09-16; First posted 2025-01-31 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Relapsed Neuroblastoma; Refractory Neuroblastoma; High-risk Neuroblastoma
Keywords: Relapsed Neuroblastoma; Refractory Neuroblastoma; High-Risk Neuroblastoma
MeSH Terms: conditions — Neuroblastoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Phase 1 Dose Escalation (Experimental): The dose escalation arm will determine the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of hALK.CAR T cells using a standard 3+3 dose escalation design.
  Interventions: Biological: Autologous hALK.CAR T cells

INTERVENTIONS:
Biological: Autologous hALK.CAR T cells — Autologous chimeric antigen receptor T cells targeting the human Anaplastic Lymphoma Kinase (ALK) receptor

SUMMARY:
This Phase 1/2 trial aims to determine the safety and feasibility of administration of autologous chimeric antigen receptor (CAR) T cells targeting the human Anaplastic Lymphoma Kinase (ALK) receptor in pediatric subjects with relapsed or refractory neuroblastoma (NB).

The trial will be conducted in two phases:

Phase 1 will determine the maximum tolerated dose (MTD) of autologous hALK.CAR T cells using a 3+3 dose escalation design. Phase 2 will be an expansion phase to determine rates of response to hALK.CAR T cells.

DETAILED DESCRIPTION:
This study consists of two phases. The primary objectives of Phase 1 and Phase 2 are:

Phase 1:

* To identify the maximum tolerated dose (MTD) of autologous hALK.CAR T cells, and the recommended phase 2 dose (RP2D) in participants with relapsed/refractory high-risk neuroblastoma.
* To evaluate the feasibility of manufacturing autologous hALK.CAR T cells.

Phase 2:

To estimate the complete response (CR) and partial response (PR) rates per revised International Neuroblastoma Response Criteria (INRC) of participants with relapsed or refractory high-risk neuroblastoma who are treated with hALK.CAR T cells.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 12 months and < 30 years at the time of consent. The first patient on each dose level will need to be age ≥ 6 years old
2. Disease Status:

   1. Patients must have histologic verification of neuroblastoma at diagnosis or at relapse
   2. Patients must have high-risk neuroblastoma according to Children's Oncology Group (COG) risk classification at time of study enrollment
   3. Patients must have persistent/refractory or relapsed disease for which standard curative measures are no longer effective, as defined in the protocol
   4. Patients must have evaluable or measurable disease per the revised International Neuroblastoma Response Criteria (INRC)
3. Adequate washout from prior treatment regimens
4. Adequate organ function
5. Adequate performance status defined as Lansky or Karnofsky performance score ≥50%
6. Subjects of reproductive potential must agree to use acceptable birth control methods
7. Signed informed consent

Exclusion Criteria:

1. Pregnant or nursing (lactating) women
2. Patients with uncontrolled active infection
3. Patients who are concurrently receiving other investigational agents
4. Patients who have received prior CART-cell or other gene-modified immune-effector cell therapy, are not eligible unless they are >8 weeks from time of infusion, have fully recovered from any associated toxicities and have documented lack of persistence of the product
5. Patients with a known additional malignancy other than non-melanomatous skin cancer or carcinoma in situ, unless not requiring active treatment and stable or disease-free for at least 3 years
6. Uncontrolled CNS metastasis
7. CNS disorder such as cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or autoimmune disease with CNS involvement which may impair the ability to evaluate neurotoxicity
8. History of severe hypersensitivity reaction to compounds used in the study
9. HIV/HBV/HCV infection
10. Patients receiving systemic steroid therapy (physiologic replacement, inhaled steroids and premedication for blood products are allowed)
11. Primary immunodeficiency or history of systemic autoimmune disease requiring systemic immunosuppression/disease modifying agents within the last 2 years
12. Uncontrolled intercurrent illness
13. Inability to comply with the study requirements

Ages: 12 Months to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-01-31 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Determine the Maximum Tolerated Dose (MTD) of hALK.CAR T cells | 5 years
  The Maximum Tolerated Dose (MTD) of hALK.CAR T cells will be determined by measuring the incidence of dose limiting toxicities (DLT) following administration of the hALK.CAR T cell product using a 3+3 dose escalation design.
Phase 1: Evaluate Manufacturing Feasibility of hALK.CAR T cells | 5 years
  Manufacturing feasibility will be evaluated as the proportion of patients undergoing leukapheresis who achieve manufacturing of a hALK.CAR T cell product that meets release criteria.
Phase 2: Estimate Response Rates | Up to 5 years
  The complete response (CR) and partial response (PR) rates per revised International Neuroblastoma Response Criteria (INRC) of subjects with relapsed or refractory high-risk neuroblastoma who are treated with hALK.CAR T cells will be estimated.

SECONDARY OUTCOMES:
Phase 1: Estimate Response Rates | 5 years
  The complete response (CR) and partial response (PR) rates per revised International Neuroblastoma Response Criteria (INRC) of subjects with relapsed or refractory high-risk neuroblastoma who are treated with hALK.CAR T cells in the Phase 1 cohort will be estimated.
Estimate Progression Free Survival and Overall Survival | 5 years
  To estimate the progression free survival (PFS) and overall survival (OS) rates of subjects with relapsed or refractory high-risk neuroblastoma who are treated with hALK.CAR T cells.
Evaluate Patient-Reported Symptoms | Up to 5 years
  Patient-reported symptoms of interest (including mood, gastrointestinal and pain symptoms) will be measured in subjects treated with hALK.CAR T cells using the Ped-PRO-CTCAE v.1 inventory prior to and until 2 years after hALK.CAR T cell infusion
Persistence of hALK.CAR T cells | Up to 5 years
  Persistence of hALK.CAR T cells will be measured by Polymerase Chain Reaction (or flow cytometry) analysis to detect and quantify survival of hALK.CAR T cells in the peripheral blood over time.
Cytokine levels in the peripheral blood | 5 years
  Activity of hALK.CAR T cells will be assessed by measuring cytokine levels in the peripheral blood over time

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Baumeister, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Boston Children's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: roberto.chiarle@childrens.harvard.edu. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu

REFERENCES:
- [Background] Bergaggio E, Tai WT, Aroldi A, Mecca C, Landoni E, Nuesch M, Mota I, Metovic J, Molinaro L, Ma L, Alvarado D, Ambrogio C, Voena C, Blasco RB, Li T, Klein D, Irvine DJ, Papotti M, Savoldo B, Dotti G, Chiarle R. ALK inhibitors increase ALK expression and sensitize neuroblastoma cells to ALK.CAR-T cells. Cancer Cell. 2023 Dec 11;41(12):2100-2116.e10. doi: 10.1016/j.ccell.2023.11.004. Epub 2023 Nov 30. PMID 38039964